CLINICAL TRIAL: NCT07035626
Title: A Trial of Spermidine for the Prevention of Radiation-Induced Xerostomia
Brief Title: A Randomized Controlled Trial of Spermidine for the Prevention of Radiation-Induced Xerostomia in Head and Neck Squamous Cell Carcinoma (Including Nasopharyngeal Carcinoma)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-2055
Record Dates: First submitted 2025-06-08; First posted 2025-06-25 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Radiation-induced Xerostomia
Keywords: Head and Neck Malignant Tumors; Radiation-induced xerostomia; Spermidine
MeSH Terms: interventions — Spermidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Cohort (Experimental): One week before the initiation of radiotherapy or concurrent chemoradiotherapy, in addition to routine health education, nursing care, and treatment, participants will start taking spermidine capsules twice daily with meals, continuing until one week after the completion of radiotherapy.
  Interventions: Drug: Spermidine
- Control Cohort (Placebo Comparator): One week before the initiation of radiotherapy or concurrent chemoradiotherapy, in addition to routine health education, nursing care, and treatment, participants will start taking placebo capsules twice daily with meals, continuing until one week after the completion of radiotherapy.
  Interventions: Drug: Spermidine simulants

INTERVENTIONS:
Drug: Spermidine — As a member of the polyamine family, spermidine is a trivalent cationic compound found in eukaryotic cells. It interacts with polyanions such as nucleic acids, proteins, and ATP through electrostatic binding, thereby maintaining genomic DNA stability, regulating gene transcription and translation, and modulating autophagy, apoptosis, oxidative stress, angiogenesis, and intercellular communication. Spermidine is indispensable for cell division and proliferation.
  Arms: Treatment Cohort
Drug: Spermidine simulants — Patients in control group were treated with Spermidine simulants, and its use method and use time are the same as intervention group.
  Arms: Control Cohort

SUMMARY:
This study is a single-center, double-blind, randomized controlled clinical trial with placebo as the control, aiming to evaluate the effectiveness of spermidine in preventing radiation-induced xerostomia during radiotherapy for head and neck tumors (including nasopharyngeal carcinoma).

DETAILED DESCRIPTION:
This study is a single-center, double-blind, randomized controlled clinical trial with placebo as the control, aiming to evaluate the effectiveness of spermidine in preventing radiation-induced xerostomia during radiotherapy for head and neck tumors (including nasopharyngeal carcinoma).

The experimental group took spermidine capsules twice a day with meals, while the placebo group took placebo capsules twice a day with meals. The appearance and taste of the placebo and spermidine were kept the same.

The primary end point was radiation-induced xerostomia, as determined by the Xerostomia Questionnaire in which a higher score indicates worse radiation-induced xerostomia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histopathologically confirmed head and neck squamous cell carcinoma (including nasopharyngeal carcinoma).
2. Aged ≥18 years and ≤80 years.
3. ECOG performance status score ≤2.
4. Receiving radical radiotherapy or concurrent chemoradiotherapy with radiation dose >50 Gy, where: Both parotid glands receive an average dose ≥25 Gy; or one gland receives a dose ≥25 Gy and the other receives any dose.
5. Blood routine parameters: hemoglobin ≥100 g/L, platelets ≥80×10⁹/L, white blood cell count ≥3.0×10⁹/L, absolute neutrophil count ≥1.5×10⁹/L.
6. Signed informed consent form.

Exclusion Criteria:

1. History of xerostomia, Sjögren's syndrome, or other known systemic diseases predisposing to dry mouth.
2. Wheat allergy or gluten intolerance.
3. Suspected or confirmed physical occlusion of bilateral salivary gland ducts.
4. Prior history of head and neck radiotherapy.
5. Use of any medications or herbal supplements that may affect salivary function within the past 30 days, or planned/final use during the study period (e.g., amifostine, cholinergic agonists [pilocarpine, cevimeline], certain β-adrenergic antagonists, anticholinergic drugs, or other known salivary function modifiers). If using saliva substitutes, patients must abstain from use for at least 24 hours prior to saliva and questionnaire data collection.
6. Poor oral hygiene or severe periodontitis.
7. Poor compliance.
8. Pregnant or breastfeeding.
9. Other patients deemed unsuitable by the investigator (e.g., concurrent severe comorbidities, mental disability, or severe emotional/psychiatric disorders).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
Radiation-induced xerostomia | Radiation-induced xerostomia will be assessed weekly from the start of radiotherapy to 3 months after its completion, totaling approximately 18-19 weeks.
  The primary end point was radiation-induced xerostomia, as determined by the Xerostomia Questionnaire in which a higher score indicates worse radiation-induced xerostomia .

SECONDARY OUTCOMES:
Unstimulated salivary flow rate | Radiation-induced xerostomia will be assessed weekly from the start of radiotherapy to 3 months after its completion, totaling approximately 18-19 weeks.
  The assessment method for unstimulated salivary flow rate is the average secretion of unstimulated saliva over 5 minutes, measured in milliliters per minute.
Quality of life (EORTC QLQ-C30) | 1 week before radiotherapy ; at the middle of radiotherapy (3 weeks after the start of radiotherapy) ; at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks) ; and 1, 2, 3 months after the end of radiotherapy.
  Quality of life will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality-of-life Questionnaire Core 30 (EORTC QLQ-C30)
Quality of life (EORTC QLQ-H&N35) | 1 week before radiotherapy ; at the middle of radiotherapy (3 weeks after the start of radiotherapy) ; at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks) ; and 1, 2, 3 months after the end of radiotherapy.
  Quality of life will be assessed using the Head and Neck Cancer Module (EORTC QLQ-H&N35).

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No